CLINICAL TRIAL: NCT00887146
Title: Phase III Intergroup Study of Radiotherapy With Concomitant and Adjuvant Temozolomide Versus Radiotherapy With Adjuvant PCV Chemotherapy in Patients With 1p/19q Co-deleted Anaplastic Glioma or Low Grade Glioma
Brief Title: Radiation Therapy With Concomitant and Adjuvant Temozolomide Versus Radiation Therapy With Adjuvant PCV Chemotherapy in Patients With Anaplastic Glioma or Low Grade Glioma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); European Organisation for Research and Treatment Center (EORTC) (Unknown); Canadian Cancer Trials Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N0577; NCI-2011-01915 (Registry Identifier: CTRP (Clinical Trials Reporting System)); EORTC-26081-22086; EudraCT-2008-007295-14; CDR0000640442 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2009-04-22; First posted 2009-04-23 (Estimated); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult anaplastic astrocytoma; adult anaplastic oligodendroglioma; adult mixed glioma
MeSH Terms: conditions — Central Nervous System Neoplasms; Astrocytoma; Oligodendroglioma; Glioma | interventions — Radiotherapy; Procarbazine; Lomustine; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (RT, procarbazine, lomustine, vincristine) (Experimental): Patients undergo 3D-CRT or IMRT on days 1-5 for 5-7 weeks. Patients also receive procarbazine hydrochloride PO on days 8-21, lomustine PO on day 1 and vincristine sulfate IV on days 8 and 29 of courses 3-8. Treatment repeats every 6-7 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: radiotherapy; Drug: procarbazine; Drug: CCNU; Drug: vincristine
- Arm B (RT, temozolomide) (Experimental): Patients undergo RT as in arm I and receive temozolomide PO QD on days 1-5 for 5-7 weeks. Beginning 4 weeks after completion of concurrent chemoradiotherapy, patients receive adjuvant temozolomide PO QD days 1-5. Treatment with adjuvant temozolomide repeats every 4 weeks for 6-12 courses in the absence of disease progression and unacceptable toxicity.
  Interventions: Drug: concomitant temozolomide (TMZ); Radiation: radiotherapy; Drug: adjuvant temozolomide (TMZ)

INTERVENTIONS:
Drug: concomitant temozolomide (TMZ) — 75 mg/m^2, orally daily
  Arms: Arm B (RT, temozolomide)
Radiation: radiotherapy
Drug: procarbazine — Days 8-21: 60 mg/m^2 orally
  Arms: Arm A (RT, procarbazine, lomustine, vincristine)
Drug: adjuvant temozolomide (TMZ) — 150 or 200 mg/m^2 orally
  Arms: Arm B (RT, temozolomide)
Drug: CCNU — Day 1: 110 mg/m^2 orally
  Arms: Arm A (RT, procarbazine, lomustine, vincristine)
Drug: vincristine — Days 8 and 29: 1.4 mg/m^2 IV
  Arms: Arm A (RT, procarbazine, lomustine, vincristine)

SUMMARY:
Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. It is not yet known whether giving radiation with concomitant and adjuvant temozolomide versus radiation with adjuvant PCV is more effective in treating anaplastic glioma or low grade glioma.

DETAILED DESCRIPTION:
This study will be a randomized phase III for patients with newly diagnosed co-deleted 1p/19q anaplastic glioma or high risk low grade glioma. The trial will only enroll patients with 1p/19q co-deletion. This study includes two arms as described in the "Arms" section. A dynamic allocation procedure will be used to allocate an equal number of patients to different arms (Arms A:B = 1:1). This procedure will balance the marginal distributions of the stratification factors among arms. The stratification factors that will be used are cooperative groups (EORTC vs. all North American groups), age (≤ 50 vs. > 50), performance score (ECOG 0-1 vs. 2), and tumor grade (anaplastic glioma vs. low grade glioma).

The primary goal is to determine whether patients who receive radiotherapy with concomitant temozolomide (TMZ) followed by adjuvant temozolomide (RT + TMZ --> TMZ) (Arm B) have a marginally better progression free survival (PFS) as compared with patients who receive radiotherapy followed by PCV chemotherapy (RT --> PCV)(Arm A).

Secondary Goals:

1. Time to Progression - To determine whether patients who receive (RT + TMZ --> TMZ) have a significantly longer time to progression (clinical or radiographic progression) as compared with patients who receive radiotherapy followed by adjuvant PCV chemotherapy (RT --> PCV).
2. Correlation between exploratory biomarkers and survival - To determine whether there is a difference in survival based on t(1;19)(q10, p10) translocation status and MGMT promoter hypermethylation status.
3. Descriptive Comparisons of Additional Secondary Endpoints - To perform descriptive comparisons of additional secondary outcome endpoints, including overall survival, objective tumor response, prognostic factor analysis and quality of life.
4. Toxicity - To determine the toxicity of the treatment in each arm and perform descriptive comparisons.
5. Neurocognitive and Quality of Life (QOL) Effects - To determine the neurocognitive and QOL effects in patients treated on this protocol and correlate these results with outcome endpoints.
6. Banking of Biospecimens and Neuroimaging Studies - To store blood products (i.e., plasma, DNA and buffy coat), tumor tissue and MRI/CT images for future scientific investigations.

After completion of study treatment, patients are followed every 12 weeks for 1 year, then every 4 months for 2 years and then every 6 months until progressive disease or until the end of study participation.

ELIGIBILITY:
Pre-Registration Inclusion Criteria:

* United States (US) and Canadian sites:

  * This review is mandatory prior to registration to confirm eligibility; patients must be willing to submit tissue samples for mandatory central pathology review submission; it should be initiated as soon after surgery as possible
* Tissue must have been determined to have local 1p/9q co-deletion and IDH mutation prior to submission for central path review

  * Tumor tissue must show co-deletion of chromosomes 1p and 19q; for eligibility, the 1p/19q analysis results will be accepted from the local site, as determined by either a locally available or reference laboratory (for US, must be Clinical Laboratory Improvement Act [CLIA] certified); acceptable methods for determination of 1p/19q loss include fluorescent in-situ hybridization (FISH), by genomic sequencing or methylomic analyses; US and Canadian sites must send a copy of the official report to the pathology coordinator and quality assurance specialist (QAS)
  * Tumor must also show evidence of IDH mutation by immunohistochemistry or genomic analyses; this should be performed at the local site (US: performed in a CLIA certified laboratory); the site must send a copy of the official report to the pathology coordinator and QAS

Registration Inclusion Criteria:

* Newly diagnosed and =< 3 months from surgical diagnosis; patients are also eligible if they have had a prior surgical procedure > 3 months earlier for low grade glioma, as long as the patient has not received prior radiation or prior chemotherapy
* Histological evidence of World Health Organization (WHO) grade III anaplastic glioma or WHO grade II low grade glioma with locally diagnosed combined 1p/19q loss and the presence of an either IDH1 or IDH2, both as established by a local or referenced laboratory qualified for the study

  * Note: mixed gliomas are eligible, regardless of the degree of astrocytic or oligodendrocytic predominance, as long as the tumor is also co-deleted for 1p and 19q
* Patients with codeleted low grade gliomas must also be considered "high risk" by exhibiting one or more of the following characteristics:

  * Age >= 40 and any surgical therapy
  * Age < 40 with prior and subtotal resection or biopsy (i.e., anything less than gross total resection)
  * Documented growth following prior surgery (NOTE: patients with prior surgery cannot have received prior radiation, chemotherapy or targeted therapy)
  * Intractable seizures
* Surgery (partial or gross total resection or biopsy) must be performed >= 2 weeks prior to registration; patient must have recovered adequately from the effects of surgery
* Absolute neutrophil count (ANC) >= 1,500/mm^3 obtained =< 21 days prior to registration
* Platelet (PLTs) count >= 100,000/mm^3 obtained =< 21 days prior to registration
* Hemoglobin (Hgb) > 9.0 g/dL obtained =< 21 days prior to registration
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) obtained =< 21 days prior to registration
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) =< 3 x ULN obtained =< 21 days prior to registration
* Creatinine =< 1.5 x ULN obtained =< 21 days prior to registration
* Negative serum or urine pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Willingness and ability to personally complete neurocognitive testing (without assistance) and willingness to complete the QOL testing, (either personally or with assistance)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0, 1 or 2
* Written informed consent
* Willingness to return to enrolling institution for follow-up during the active monitoring phase (that is, the active treatment and observation portion) of the study); patients who have been formally transferred to another active and approved site participating in this study would not need to return to the enrolling institution for this purpose
* Willingness to allow the provision of tissue samples for correlative research, as long as adequate tissues are available; patients will not be excluded from participation in the study, if they are willing to allow provision of tissues for the correlative research, but there are insufficient quantities of tissue for the correlative analyses (e.g., a patient otherwise eligible and willing who had biopsy only) Willingness to allow the provision of blood samples for correlative research; patients are not excluded from participation in the study, if they are willing to provide the mandatory biospecimens for translational/correlative research, but for logistical reasons the specimens(s) were not obtainable or if the volume collected was insufficient

Registration Exclusion Criteria:

* The following categories are ineligible:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception or contraceptive method during this study and 6 months following the completion of chemotherapy treatments
* History of prior radiation therapy or chemotherapy for glioma; note: patients who have a history of prior low grade glioma (with or without a distant history of prior surgery for that glioma), but who have never received prior chemotherapy or radiation therapy for the glioma are eligible for the study
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Concomitant serious immunocompromised status (other than that related to concomitant steroids) that would compromise the safety of the patient on the study
* Patients known to be human immunodeficiency virus (HIV) positive and currently receiving retroviral therapy are not eligible; note: patients known to be HIV positive, but without clinical evidence of an immunocompromised state, are eligible for the study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Receiving any other investigational agent that would be considered as a treatment for the primary neoplasm
* Other active malignancy within 5 years of registration; exceptions: non-melanotic skin cancer or carcinoma-in-situ of the cervix; note: if there is a history of prior malignancy, the patient is not eligible if they are receiving other specific treatment (with the exclusion of hormonal therapy or Her-2 inhibitors) for their cancer or if they have received prior total body irradiation which included the brain
* History of myocardial infarction =< 6 months, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* Recent history of hepatitis infection or if the treating physician determined that the patient would be at significant risk of reactivation of hepatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2029-10-31 (Estimated); Study Completion 2029-10-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | Time from study registration to time of tumor progression or death due to any cause, whichever comes first, assessed up to 16 years
  The distribution of progression free survival for Arms A and B will be estimated using the Kaplan-Meier method. The hazard ratios and median progression free survival (PFS) will be estimated with their confidence intervals. The Cox proportional hazards model will be used to assess whether the distributions of progression survival times differ with respect to treatment regimen having adjusted for all stratification factors (cooperative groups, age, and performance score). Both non-inferiority and superiority will be tested in this trial for the primary goal and no multiple-comparison adjustment will be considered.

SECONDARY OUTCOMES:
Time to progression | Time from study registration to the earliest evidence of clinical progression, radiographic progression or neurocognitive progression, assessed up to 16 years
  Estimated by Kaplan-Meier method and analyzed by Cox regression model adjusting all stratification factors. Correlations among baseline neurocognitive test scores and progression free survival will be analyzed using Cox proportional hazards model.
Time to neurocognitive progression, assessed using the Hopkins Verbal Learning Test-Revised for Free Recall, Delayed Recall, and Delayed Recognition; the Controlled Oral Word Association test; and the Trail Making Test Part A or B | Time from study registration to the first cognitive failure, assessed up to 16 years
  Estimated by Kaplan-Meier method and analyzed by Cox regression model adjusting all stratification factors. For each test in the battery, a standard error of measurement will be used to derive the Reliable Change Index (RCI) which will be used to represent the 90% confidence interval for the difference in raw scores from baseline to follow-up assessment will be coded as 1 (deterioration), 2 (no change), and 3 (improved) according to the RCI.
Overall survival | Time from study registration to time of death due to any cause, assessed up to 16 years
  The Cox proportional hazards model will be used to assess whether the distributions of overall survival times differ with respect to treatment regimen having adjusted for all stratification factors (cooperative groups, age, and Performance Score). The distribution of overall survival for Arm A and B will be estimated using the Kaplan-Meier method. The hazard ratios and median survivals will be estimated with their 95% confidence intervals.
Objective tumor response defined as a complete response or partial response | Up to 16 years
  Summarized for each arm and compared between the arms using the Chi square test.
Treatment-related adverse events according to National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | Up to 16 years
  The maximum grade for each type of treatment-related adverse event will be recorded for each patient, and frequency tables for each arm will be reviewed to determine patterns. In addition, will review all adverse event data that is graded as 3, 4, or 5 and classified as either "unrelated" or "unlikely to be related" to study treatment in the event of an actual relationship developing. Adverse events and treatment-related adverse events will be evaluated using all patients. Treatment-related adverse events will be tabulated for each arm.

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Jaeckle, MD, Study Chair — Mayo Clinic
Locations (291):
- United States (271):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Providence Hospital, Mobile, Alabama
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Saint Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Arizona Oncology-Deer Valley Center, Phoenix, Arizona
  - Arizona Oncology Services Foundation, Scottsdale, Arizona
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Community Cancer Institute, Clovis, California
  - University Oncology Associates, Clovis, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Kaiser Permanente-Ontario, Ontario, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Sutter Cancer Centers Radiation Oncology Services-Vacaville, Vacaville, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - The Medical Center of Aurora, Aurora, Colorado
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Saint Francis Cancer Center, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Banner McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Yale University, New Haven, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Emory Proton Therapy Center, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - AMITA Health Adventist Medical Center, La Grange, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - McFarland Clinic - Ames, Ames, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Mission Cancer and Blood - West Des Moines, Clive, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Mission Cancer and Blood - Des Moines, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Mission Cancer and Blood - Laurel, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Hospital Pavilion and Medical Campus, Louisville, Kentucky
  - Norton Brownsboro Hospital and Medical Campus, Louisville, Kentucky
  - West Jefferson Medical Center, Marrero, Louisiana
  - Maine Medical Center-Bramhall Campus, Portland, Maine
  - Maine Medical Center- Scarborough Campus, Scarborough, Maine
  - Maine Medical Partners Neurology, Scarborough, Maine
  - Maine Medical Partners - South Portland, South Portland, Maine
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Cancer Trials Support Unit, Rockville, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Hematology and Oncology, Lincoln, Nebraska
  - Cancer Partners of Nebraska, Lincoln, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Nebraska Cancer Specialists - Omaha, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Regional West Medical Center Cancer Center, Scottsbluff, Nebraska
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - GenesisCare USA - Las Vegas, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New York-Presbyterian/Brooklyn Methodist Hospital, Brooklyn, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Highland Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Altru Cancer Center, Grand Forks, North Dakota
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Saint Luke's Hospital-Anderson Campus, Easton, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - UTMB Cancer Center at Victory Lakes, League City, Texas
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Intermountain Medical Center, Murray, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Tri-Cities Cancer Center, Kennewick, Washington
  - Skagit Regional Health Cancer Care Center, Mount Vernon, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - FHCC South Lake Union, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
- Medical University Vienna, Vienna, Austria
- Alegemeen Ziekenhuis Middelheim, Antwerp, Belgium
- Canada (11):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - London Regional Cancer Program, London, Ontario
  - Ottawa Hospital and Cancer Center-General Campus, Ottawa, Ontario
  - Odette Cancer Centre- Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - CHUM - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
- France (3):
  - Centre Leon Berard, Lyon
  - Centre Antoine Lacassagne, Nice
  - Gustave Roussy, Villejuif
- Netherlands (4):
  - Academ Zienkenhuis Bij De University, Amsterdam
  - University Medical Center Groningen, Groningen
  - Maastro Clinic-Maastricht Radiation Oncology, Maastricht
  - Erasmus University Medical Center, Rotterdam

REFERENCES:
- [Derived] Cerhan JH, Anderson SK, Butts AM, Porter AB, Jaeckle K, Galanis E, Brown PD. Examiner accuracy in cognitive testing in multisite brain-tumor clinical trials: an analysis from the Alliance for Clinical Trials in Oncology. Neurooncol Pract. 2019 Jul;6(4):283-288. doi: 10.1093/nop/npy048. Epub 2018 Nov 24. PMID 31386061
- [Derived] Drappatz J, Lieberman F. Chemotherapy of Oligodendrogliomas. Prog Neurol Surg. 2018;31:152-161. doi: 10.1159/000467376. Epub 2018 Jan 25. PMID 29393183
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — https://www.cancer.gov/about-cancer/treatment/clinical-trials/search/v?id=NCI-2011-01915&q=N0577